CLINICAL TRIAL: NCT01809470
Title: Metabolic Response to Playing Video Games
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UCL-VG-001
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-01

CONDITIONS: Blood Pressure
Keywords: Blood pressure; Appetite; Heart rate; Salivary cortisol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Watching TV (Experimental): Watching TV (comedy, 'Friends') for 1 hour
  Interventions: Behavioral: Watching TV
- FIFA2013 (Experimental): Playing the video game 'FIFA2013' for 1 hour
  Interventions: Behavioral: FIFA2013
- Call of Duty (Experimental): Playing the video game 'Call of duty' for 1 hour
  Interventions: Behavioral: Call of Duty

INTERVENTIONS:
Behavioral: FIFA2013 — Playing FIFA2013 for 1 hour
  Arms: FIFA2013
Behavioral: Call of Duty — Playing Call of Duty for 1 hour
  Arms: Call of Duty
Behavioral: Watching TV — Watching TV for 1 hour
  Arms: Watching TV

SUMMARY:
The study is investigating the metabolic response to playing competitive non-violent and competitive violent video games. The primary hypothesis is that the metabolic response in the violent game group will differ from the other two groups, due to activation of the stress response. The investigators are using an experimental approach, whereby 72 young men are randomised to one of three groups: watching television (TV), playing the non-violent video game 'FIFA2013', or playing the violent video game 'Call of Duty'. Participants arrive fasted, and are given a standardised breakfast. After measurements of weight, height and waist girth, they then are assigned to one of the three groups. Baseline blood pressure, heart rate and appetite/mood data are collected, along with a saliva sample for measurement of the 'stress' hormone, cortisol. The investigators will collect these data again at 4 time-points during the one hour game-playing session. At the end of the study, the allow the participants half an hour of rest, during which they can choose from a variety of sweet or savoury snacks. The investigators will compare the data from the three groups, to test whether changes in blood pressure, heart rate and salivary cortisol, as well as snack consumption, are greater in the group playing the violent game.

DETAILED DESCRIPTION:
Our study is investigating the metabolic response to playing competitive non-violent and competitive violent video games. Our primary hypothesis is that the metabolic response in the violent game group will differ from the other two groups, due to activation of the stress response.

We are using an experimental approach, whereby 72 young men are randomised to one of three groups: watching TV, playing the non-violent video game 'FIFA2013', or playing the violent video game 'Call of Duty'. All participants must already have some experience playing the two games, so that whichever group they are assigned to, they can comply with the protocol.

Participants arrive after an overnight fast, and are given a standardised breakfast (a muffin, approx 300 kcal, and a glass of water). After measurements of weight, height and waist girth, they then are assigned to one of the three groups, and allowed to familiarise themselves with the games console or TV. Baseline data on blood pressure (in triplicate, Accutor digital monitor), heart rate (Polar monitor) and appetite/mood (visual analogue scale) are collected, along with a saliva sample for measurement of the 'stress' hormone, cortisol, as well as satiety hormones sich as leptin and ghrelin. We will collect these data again at 4 time-points during the one hour game-playing session, by pausing the game or TV for 4 minutes at 15, 30, 45 and 60 minutes after the session starts.

At the end of the study, we allow the participants half an hour of rest, during which they can choose from a variety of sweet or savoury snacks or fruit, and several drinks.

We will compare the data from the three groups, to test whether changes in blood pressure, heart rate, appetite/mood and salivary hormones, as well as snack consumption, are greater in the group playing the violent game.

ELIGIBILITY:
Inclusion Criteria:

* BMI >25 kg/m2

Exclusion Criteria:

* smoker
* weight change >3 kg in the previous three months
* psychiatric disorder
* uncontrolled hypertension
* coronary heart disease, heart failure and central or peripheral arteriopathies
* alcohol consumption > 21 units/week.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Over the 90 minutes of the study
  Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Heart rate | Over the 90 minute duration of the study
  Heart rate by Polar monitor
Appetite | Over the 90 minute duration of the study
  Appetite by visual analogue scale, and by a test meal at the end of the study
Stress | Over the 90 minute duration of the study
  Salivary cortisol
Satiety | Over the 90 minute duration of the study
  Salivary ghrelin and leptin

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Wells, PhD, Principal Investigator — UCL Institute of Child Health
Locations (1):
- UCL Institute of Child Health, London, United Kingdom